CLINICAL TRIAL: NCT07142473
Title: Mastocytosis From Pediatric Age to Adulthood: Local Registry of Cutaneous and Systemic Mastocytosis
Acronym: MaRe
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Valeria Brazzelli, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: MaRe
Record Dates: First submitted 2025-02-17; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-02

CONDITIONS: Cutaneous Mastocytosis; Systemic Mastocytosis
MeSH Terms: conditions — Mastocytosis, Cutaneous; Mastocytosis, Systemic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients diagnosed with cutaneous or systemic mastocytosis

SUMMARY:
Given the renewed focus on mastocytosis (recognized in Italy as a rare disease since 2018) and emerging clinical and immunogenetic knowledge, and considering the rarity of the disease and limited understanding of its progression, this observational study aims to analyze epidemiological, clinical, genetic, immunohistochemical, and laboratory characteristics of patients with mastocytosis. This will help expand knowledge about the disease and identify prognostic variables useful in developing a personalized therapeutic approach.

This registry aims to collect retrospective and prospective data on patients with cutaneous and systemic mastocytosis attending the Dermatology Unit at the IRCCS Fondazione Policlinico San Matteo.

This is a single-center longitudinal hospital registry including patients with cutaneous and systemic mastocytosis, collected retrospectively and prospectively to assess the clinical, serological, hematological, and molecular characteristics of patients with cutaneous and systemic mastocytosis and their correlation with specific outcomes such as disease variant (cutaneous or systemic), extent of skin involvement, and survival rate.

ELIGIBILITY:
Inclusion criteria:

- Cutaneous or systemic mastocytosis diagnosys attending the Dermatology Outpatient Clinics of the UOC Dermatology Unit Fondazione IRCCS Policlinico San Matteo

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed with cutaneous or systemic mastocytosis attending the Dermatology Outpatient Clinics of the UOC Dermatology Unit Fondazione Policlinico San Matteo IRCCS Pavia will be eligible for inclusion in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2034-01-26 (Estimated); Study Completion 2034-01-26 (Estimated)

PRIMARY OUTCOMES:
Prevalence of the systemic disease variant in the examined population | January 2034
  The prevalence and the 95% exact binomial confidence interval will be presented

SECONDARY OUTCOMES:
Association between clinical, serological, hematological, and molecular characteristics and the disease variant (cutaneous or systemic) | January 2034
  The association will be evaluated using a multivariate logistic model; the number of covariates will be limited by the number of systemic mastocytosis cases, maintaining a 1:10 ratio. The selection of covariates will be made a priori based on scientific knowledge. Odds ratios (OR) and their corresponding 95% confidence intervals (CI) will be reported. The model's discriminatory ability (area under the ROC curve) and its calibration (graphically) will be calculated
Association between family history and age of disease onset | January 2034
  The analysis will be performed using a multivariate logistic model
Survival rate in relation to the disease variant (cutaneous or systemic) | January 2034
  The survival rate will be reported as deaths per 100 person-years; the start date for follow-up will be the diagnosis of the disease. The groups will be compared using the log-rank test, and survival will be described using Kaplan-Meier curves. A Cox model will be used to derive the hazard ratio (HR) and the corresponding 95% confidence interval (CI). Harrell's C-statistic will be calculated to assess the model's discriminatory ability. Estimates will be adjusted, where possible, for potential confounding factors
Association between c-KIT mutation in blood and clinical characteristics of the patient | January 2034
  The analysis will be performed using a multivariate logistic model
Evaluation of dermatoscopic characteristics in relation to the clinical presentation of the disease and the patient's age | January 2034
  The analysis will be performed using a multivariate logistic model. For the purposes of the analysis, age will be dichotomized at the median. Linear regression models may also be used

CONTACTS AND LOCATIONS:
Locations (1):
- SC Dermatologia, Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No